CLINICAL TRIAL: NCT04957485
Title: A Phase 1, Open-Label (JYNNEOS®), Double-Blind (TPOXX® And Placebo), Multicenter, Randomized, Placebo-Controlled, Drug-Vaccine Interaction Study To Evaluate the Impact of TPOXX on JYNNEOS Immunogenicity
Brief Title: Study to Assess the Safety and Immunogenicity of TPOXX® When Administered Orally for 28 Days With JYNNEOS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SIGA Technologies (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIGA-246-028
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — tecovirimat; Smallpox Vaccine; smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- JYNNEOS + TPOXX (Active Comparator): An oral dose of 600 mg (3 × 200 mg capsules) TPOXX BID (every 12 hours [±30 minutes]) for 28 days and a single AM SC dose of 0.5 mL JYNNEOS on Day 1 and Day 29. JYNNEOS will be administered with TPOXX concomitantly on Day 1
  Interventions: Drug: Tecovirimat; Drug: Smallpox and Mpox Vaccine
- JYNNEOS + matching TPOXX placebo (Placebo Comparator): An oral dose of placebo (3 capsules identical to TPOXX) BID (every 12 hours [±30 minutes]) for 28 days and a single AM SC dose of 0.5 mL JYNNEOS on Day 1 and Day 29. JYNNEOS will be administered with TPOXX placebo concomitantly on Day 1.
  Interventions: Drug: Smallpox and Mpox Vaccine; Other: Placebo

INTERVENTIONS:
Drug: Tecovirimat — oral antiviral
  Other Names: TPOXX
  Arms: JYNNEOS + TPOXX
Drug: Smallpox and Mpox Vaccine — vaccine
  Other Names: JYNNEOS
Other: Placebo — TPOXX Placebo
  Arms: JYNNEOS + matching TPOXX placebo

SUMMARY:
This study is designed to evaluate the immunogenicity profile of JYNNEOS® when 2 doses are administered subcutaneously (SC) 4 weeks apart; and potential immunological interference while concomitantly administering TPOXX or placebo orally twice daily (BID) for 28 days.

DETAILED DESCRIPTION:
This is a Phase 2, open-label (JYNNEOS), double-blind (TPOXX and placebo), multicenter, randomized, placebo-controlled, drug-vaccine interaction study to examine whether administering TPOXX with JYNNEOS concomitantly affects JYNNEOS immunogenicity in healthy adult subjects. A total of 100 subjects (approximately 50 subjects per treatment group), ages 18 to 42, inclusive, will be enrolled and randomly assigned to 1 of 2 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Subject is a healthy male or female between 18 and 42 years of age, inclusive, at the time of informed consent.
2. Subject has a resting heart rate >40 beats per minute (bpm) or <110 bpm at screening.
3. Subject has negative test for HIV antibodies, hepatitis B surface antigen, and hepatitis C virus antibody.
4. Subject has white blood cells ≥2500/mm3 and <11,000/mm3.
5. Subject has hemoglobin within normal limits.
6. Subject has platelets ≥ lower normal limits.
7. Subject has adequate renal function defined as a calculated creatinine clearance >60 mL/min as estimated by the Cockcroft-Gault equation.
8. Creatinine in males ≤1.7 mg/dL and in females ≤1.4 mg/dL (1.3 times the upper laboratory reference range).
9. Subject has adequate hepatic function in the absence of other evidence of significant liver disease defined as:

   1. Total bilirubin <1.5 times above the upper laboratory reference range
   2. Alanine aminotransferase <1.5 times above the upper laboratory reference range
   3. Aspartate aminotransferase <1.5 times above the upper laboratory reference range
   4. Alkaline phosphatase <1.5 times above the upper laboratory reference range.
10. Male subject has a QT interval corrected using Fridericia's formula (QTcF) <450 ms or female subject has a QTcF <470 ms at screening or Day 1.
11. Women of childbearing potential have a negative B-human chorionic gonadotropin pregnancy test (serum) at the screening visit and a negative urine pregnancy test on Day 1 before receipt of study drug, and meet one of the following criteria:

    1. The subject or their partner has undergone surgical sterilization.
    2. The subject is postmenopausal, defined as 12 consecutive months with no menses without an alternative medical cause and has a documented plasma follicle stimulating hormone level >40 mIU/mL.
    3. The subject agrees to be abstinent (heterosexually inactive) for the duration of the study.
    4. The subject agrees to consistently use one of the following methods of contraception from the beginning of screening (which they had been consistently using for at least 30 days before the first dose of study drug) through 30 days after the second JYNNEOS injection:

    i. Condoms, male or female, with a spermicide NOTE: For male subjects, condoms must be used for 90 days after the second JYNNEOS injection. Male and female condoms should not be used together, as this can reduce their effectiveness.

    ii. Diaphragm or cervical cap with spermicide iii. Intrauterine device with spermicide iv. Oral contraceptives or other hormonal methods NOTE: Another nonhormonal method of contraception must be used in conjunction with oral contraceptives.

    v. Male sexual partner who had undergone a vasectomy at least 3 months before screening.
12. Male subjects must agree to not donate sperm from the first JYNNEOS injection through 90 days after the second JYNNEOS injection.
13. The subject agrees to not donate blood or blood components for 4 weeks after the completion of the study.
14. The subject agrees to not consume caffeine- or xanthine-containing products during all study visits; sodas, coffee, and tea designated as caffeine-free or noncaffeinated may be consumed on study days; caffeine may be consumed while at home and between study visits.
15. The subject agrees to comply with the study dietary requirements.
16. The subject agrees to comply with all protocol requirements.
17. The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening.
18. The subject has read, signed, and dated the informed consent, having been advised of the risks and benefits of the trial in a language understood by the subject and prior to performance of any trial-specific procedure.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Subject is a female who is pregnant or breastfeeding or planning to become pregnant within 3 months after the second JYNNEOS injection.
2. Subject has a history or suspected exposure of smallpox, monkeypox or cowpox disease, or previous vaccination with any poxvirus-based vaccine.
3. Subject has received any vaccinations within 28 days prior to Day 1 or plans to receive a vaccination at any time during the treatment period or within 28 days after Day 29.
4. Subject weighs 120 kg or more.
5. Subject has been administered or plans to be administered immunoglobulins and/or any blood products during a period starting from 3 months prior to administration of the vaccine and ending at trial conclusion.
6. Subject has used any investigational or nonregistered drug or vaccine other than the trial vaccines within 28 days preceding the first dose of the trial vaccine or planned administration of such a drug /vaccine during the trial period, including the COVID-19 vaccine prior to marketing approval by the FDA.
7. Subject has a known or suspected history of smallpox vaccination defined as visible vaccination scar or documentation of smallpox vaccination or as reported by the subject.
8. Subject has had a previous anaphylactic reaction, severe systemic response, or serious hypersensitivity to a prior immunization.
9. Subject has a history of any clinically significant conditions including the following:

   * Asthma treated with oral systemic steroids within the past 6 months
   * Diabetes mellitus (type 1 or 2), with the exception of gestational diabetes
   * Hypertension that is poorly controlled (repeat readings >140 mm Hg systolic and/or >90 mm Hg diastolic)
   * Serious angioedema episodes within the previous 3 years or requiring medication in the previous 2 years
   * Head trauma resulting in a diagnosis of traumatic brain injury other than concussion
   * Frequent episodes of headache
   * Active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded
   * History of or active immunodeficiency or immunosuppression caused by acquired or congenital diseases or caused by ongoing treatments such as chronic (greater than 14 days) high-dose corticosteroids (smaller than 5 mg prednisone [or equivalent] per day applied systemically, i.e., parenterally or orally), chronic or planned treatment with steroid eye drops or ointment at time of enrollment or radiation, or immunosuppressive drugs; low-dose corticosteroid topical products and nasal sprays used sporadically, i.e., pro re nata (according to circumstances) are permissible
10. Subject has received treatment in another clinical study of an investigational drug (or medical device) or investigational vaccine within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug.
11. Subject has previously participated in this or any other clinical trial involving TPOXX (tecovirimat).
12. Subject has known allergies to any components or excipients of TPOXX or JYNNEOS.
13. Subject has any condition possibly affecting drug absorption (e.g., previous surgery on the gastrointestinal tract, including removal of parts of the stomach, bowel, liver, gallbladder, or pancreas, with the exception of appendectomy).
14. Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of the first JYNNEOS injection), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease. Exceptions to these criteria (e.g., stable, mild joint disease unassociated with collagen vascular disease) may be made following discussions with the medical monitor.
15. Subject has a history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, chest pain (that is diagnosed as cardiac related) or trouble breathing on exertion, or risk factors for torsades de pointes (e.g., heart failure, hypokalemia).
16. Subject has a blood pressure considered to be clinically significant by the investigator. Blood pressure may be retested twice in the sitting position at 5-minute intervals.
17. Subject has a family history of an immediate family member (father, mother, brother, or sister) who has had an onset of ischemic heart disease before the age of 50 years.
18. Subject is 20 years of age and older and has a ≥10% risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's Risk Assessment Tool: https://www.mcw.edu/calculators/ldl-cholesterol-goal-level.
19. Subject has a seizure disorder or history of seizures (does not include childhood febrile seizures) or a past history that increases seizure risks such as significant head injury that caused loss of consciousness or other changes in the subject's daily function, concussion, stroke, central nervous system infection or disease, or alcohol or drug abuse or family history of idiopathic seizures.
20. Subject has a history of a peptic ulcer or significant gastrointestinal bleeding.
21. Subject has had radiation or x-ray treatment (not routine x-rays) within the last 3 months.
22. Subject is post organ and bone-marrow transplant whether or not receiving chronic immunosuppressive therapy.
23. Subject has a bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with blood draws.
24. Subject has neutropenia or other blood dyscrasia determined to be clinically significant by the investigator.
25. Subject has a major congenital defects or serious chronic illness, including any cancer other than the following: a) any nonmetastatic cancer (excluding hematologic malignancies) or melanoma of which the participant has been disease-free for at least 5 years and b) localized skin cancer, resected (including squamous cell and basal cell carcinomas).
26. Subject has active or a history of chronic alcohol abuse and/or intravenous and/or nasal drug abuse (within the past 6 months).
27. Subject has a current or recent (<30 days before screening) history of clinically significant bacterial, fungal, or mycobacterial infection.
28. Subject has a known clinically significant chronic viral infection (e.g., human T-cell lymphotropic virus I or II) or acute disease (illness without fever) at the time of enrollment. Note that screening laboratory tests may be delayed allowing the resolution of a transient acute condition or the subject may be rescreened.
29. Subject has any confirmed or suspected immunodeficiency condition (congenital or secondary) or autoimmune disease based on medical history and physical examination, e.g., Guillain Barré.
30. Subject has a family history of congenital or hereditary immunodeficiency.
31. Subject has any planned elective surgery during the study through 12 months after the last vaccination.
32. Subject has planned receipt of immunoglobulins and/or any blood products within the 3 months preceding study enrollment or at any point during the study period until after the final safety telephone contact.
33. Subject is a member or family member of the investigator site team.
34. Subject demonstrates long-term use (≥14 consecutive days) of glucocorticoids, including oral or parenteral prednisone or equivalent (>20 mg total dose per day), or high-dose inhaled steroids (>800 µg/day of beclomethasone dipropionate or equivalent) within the preceding 30 days (low-dose [≤800 µg/day of beclomethasone dipropionate or equivalent] inhaled and topical steroids are allowed).
35. Subject has donated >450 mL blood or blood components within 30 days before the first dose of study drug.
36. Subject reports participation in strenuous activity or contact sports within 24 hours before the first dose of study drug.
37. Subject has a positive test result for amphetamines (including methamphetamines and ecstasy/methylenedioxymethamphetamine), barbiturates, benzodiazepines, cannabinoids (including tetrahydrocannabinol), cocaine metabolites, opiates (including heroin, codeine, and oxycodone), or alcohol at screening or Day 1.
38. Subject has used any of the following prohibited medications within 14 days (or 5 half lives, whichever is longer) before the first JYNNEOS injection: antidiabetic medication; anticoagulants; anticonvulsants; substrates of the breast cancer resistance protein transporter including methotrexate, mitoxantrone, imatinib, irinotecan, lapatinib, rosuvastatin, sulfasalazine, and topotecan; substrates of CYP2C8 including repaglinide, paclitaxel, montelukast, pioglitazone, rosiglitazone; and substrates of CYP2C19 including S-mephenytoin, clobazam, diazepam, rabeprazole, voriconazole, lansoprazole, and omeprazole. Medications not listed here that are known (or thought) to be CYP3A4 substrates may be allowed at the investigator's discretion, after consultation with the medical monitor, if administration poses little to no risk to the subject.
39. Subject has used any prescription antiviral drugs with the intention of COVID-19 prophylaxis, including those that are thought to be effective for prevention of COVID-19 but have not been licensed for this indication, within 1 month prior to study entry or during the study.
40. In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 59 Days
  Number of participants with adverse events when TPOXX or TPOXX Placebo is coadministered with JYNNEOS
Immunogenicity | Day 43
  Least squared geometric mean

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hruby, Ph.D., Study Director — SIGA Technologies
Locations (2):
- United States (2):
  - Meridian Clinical Research, Omaha, Nebraska
  - Aventiv Research Inc, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No